CLINICAL TRIAL: NCT06407908
Title: Urdu Translation and Psychoprometric Properties Of Pediatric Version Of Eating Assessment Tool
Brief Title: Urdu Translation Of Pediatric Version Of Eating Assessment Tool
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/23/0788
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: validation; translation; eating disorder; PEDI-EAT-10
MeSH Terms: conditions — Cerebral Palsy; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dysphagia encompasses challenges encountered during the many stages of swallowing, including the oral phase, commencement of the swallow, pharyngeal phase, and esophageal phase. The incidence of pediatric dysphagia is on the rise as a result of advancements in medical care that have led to higher survival rates among infants born prematurely, with low birth weight, and with complex medical disorders. The Eating Assessment Tool (EAT-10), consisting of 10 items, was first developed for infant patients.

(PEDI-EAT-10) will be translated into Urdu language by using forward backwards translation method. Two bilingual speakers expert in both Urdu and English languages will assist the researcher in the forward translation of the tool. This final translated version will be then tested for validity and reliability on all participants of the study. The psychometric properties of the tool will be assessed including reliability, internal consistency, and item discrimination.

DETAILED DESCRIPTION:
A mix method approach will be applied

1. Forward translation
2. Reconciliation of items
3. Backward translation
4. Review of forward and backward translation
5. Pre-testing (cognitive interviewing)
6. Validation study The process of translation followed the guidelines in the translation manual. Translators translate the pediatric version of eating assessment tool (Pedi-EAT-10), independently from each other into the Urdu language considering the following guidelines: using natural language acceptable to the broader public, performing a clear, simple, and understandable translation, avoiding lengthy and complicated sentences. This will be followed by a backward translation to ensure that the content, from the conceptual point of view, had not been modified in the translation. A native English translator was requested to carry out the back-translation, and all discrepancies were identified and corrected. To show whether all items are easily understood and acceptable to the patients, pretesting the final translated questionnaire will be conducted by administering it to patients with a varying education level. The questions that were not easily understood were discussed and redrafted by a panel of researchers until all interviewees understood all items.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children diagnosed with eating disorders
* Age from 3 to 15 years

Exclusion Criteria:

* Parents with children Unable to understand the questionnaire
* Parents with children who have Intellectual disability and any organic type of incontinence, neurological or anatomical problems
* Parents with who have children Severe cognitive decline or dementia
* Parents with children cannot understand Urdu.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample size is 42.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Pediatric Version of the Eating Assessment Tool (Pedi-EAT-10) | 6 months
  This resource is essential for determining how these obstacles affect a child's health and food consumption. The pediatric version is specially designed to evaluate a child's eating and swallowing skills, taking into consideration their specific developmental and physiological needs.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Ahsan, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varni JW, Limbers CA, Neighbors K, Schulz K, Lieu JE, Heffer RW, Tuzinkiewicz K, Mangione-Smith R, Zimmerman JJ, Alonso EM. The PedsQL Infant Scales: feasibility, internal consistency reliability, and validity in healthy and ill infants. Qual Life Res. 2011 Feb;20(1):45-55. doi: 10.1007/s11136-010-9730-5. Epub 2010 Aug 22. PMID 20730626